CLINICAL TRIAL: NCT06773663
Title: Evaluation of Biodistribution, Dosimetry, Diagnostic and Surgery-guiding Ability of Al18F-NOTA-Pentixafor PET Imaging for Patients With Primary Aldosteronism: A Prospective, Single-center Study
Brief Title: Application of Al18F-NOTA-Pentixafor PET/CT for Primary Aldosteronism
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K5164
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-10

CONDITIONS: Primary Aldosteronism; Primary Aldosteronism Due to Aldosterone Producing Adenoma
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-NOTA-Pentixafor PET/CT (Experimental): Evaluation of dosimetry, safety, diagnostic accuracy, and surgical guidance ability of Al18F-NOTA-Pentixafor PET/CT in patients with primary aldosteronism
  Interventions: Combination Product: Al18F-NOTA-Pentixafor PET/CT

INTERVENTIONS:
Combination Product: Al18F-NOTA-Pentixafor PET/CT — Participants will receive an intravenous injection of Al18F-NOTA-Pentixafor, prepared on-site and measured by qualified personnel using a dose calibrator, with readings and time recorded. The radiopharmaceutical will be slowly administered through a three-way stopcock, followed by a flush with 5 mL of normal saline.
  The recommended dose is approximately 4.81 MBq/kg (0.13 mCi/kg) body weight, with variations depending on drug yield and clinical scheduling.
  CT and PET imaging are planned 45-90 minutes after administration, with adjustments based on drug yield and equipment availability.

SUMMARY:
This prospective, single-center study investigates the biodistribution, dosimetry, safety, diagnostic performance of Al18F-NOTA-Pentixafor PET imaging in patients with primary aldosteronism. And evaluates the potential of Al18F-NOTA-Pentixafor PET imaging in surgical strategy guidance.

DETAILED DESCRIPTION:
Hypertension has a high prevalence, being a leading cause of premature death in 1.4 billion adults worldwide. Primary aldosteronism (PA) is the most common cause of secondary hypertension. Guidelines recommend that 50% of people with hypertension should be screened for PA, yet fewer than 1% of PA patients have undergone screening and treatment. Aldosterone-producing adenoma (APA) and idiopathic hyperaldosteronism (IHA) are the primary subtypes of PA, accounting for approximately 35% and 60% of cases, respectively. Early diagnosis and treatment can improve prognosis and enhance patients' quality of life. Screening for PA, particularly in patients with resistant hypertension or newly diagnosed hypertension, has practical clinical significance.

Currently, adrenal vein sampling (AVS) is considered the "gold standard" for PA subtyping, allowing for the identification of unilateral dominant secretion, with a sensitivity of 95% and a specificity of 100%. However, AVS is an invasive procedure, expensive, requires hospitalization, is technically challenging, and carries risks of catheterization failure and post-procedural complications. Thus, it is difficult to implement AVS on a large scale across medical facilities. Conventional imaging techniques such as CT have low detection efficacy for small adrenal nodules, falling short of clinical diagnostic and therapeutic needs.

CXCR4 is a typical G-protein-coupled receptor primarily located on the cell membrane. Upon activation, it stimulates cell migration and activation, playing a key role in hematopoiesis, immunity, inflammation, and cancer regulation. Recent studies have found that CXCR4 is highly expressed on the cell membrane of APA and is significantly correlated with the expression level of aldosterone synthase (CYP11B2), while it is expressed at low levels in non-functional adenomas. The nuclear medicine molecular probe, 68Ga-Pentixafor, is a specific ligand for CXCR4. By specifically binding to CXCR4 receptors on the cell membrane, it provides functional imaging through PET/CT, offering a simple, direct, and effective reference for PA subtyping and clinical decision-making.

Al18F-NOTA-Pentixafor is an imaging agent targeting CXCR4, and in vitro experiments have shown its specific binding to CXCR4 with high affinity. Therefore, Al18F-NOTA-Pentixafor PET imaging can be used for the non-invasive localization of all CXCR4-positive lesions in vivo, including APA. However, currently, only limited research has investigated the application of Al18F-CXCR4 receptor imaging in PA, and no studies have yet examined its potential value for surgical guidance in patients with PA. Al18F-NOTA-Pentixafor can be synthesized automatically in large quantities within a short time. If its imaging performance is not inferior to that of 68Ga-Pentixafor, it would be more advantageous for large-scale clinical application.

This prospective, single-center study aims to assess the biodistribution, dosimetry, safety, and diagnostic efficacy of Al18F-NOTA-Pentixafor PET imaging in patients with primary aldosteronism. Furthermore, it evaluates the potential of Al18F-NOTA-Pentixafor PET imaging to guide surgical strategies for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with adrenal masses suspected to be aldosterone-producing adenomas based on routine imaging (e.g., CT scans), or clinically diagnosed primary aldosteronism patients requiring subtyping
2. Signed written informed consent, with willingness and ability to comply with study procedures.
3. Female participants must be surgically sterilized or postmenopausal for over a year; if not, reliable contraception is required.
4. Male participants must use reliable contraception during the study and refrain from sperm donation.

Exclusion Criteria:

1. Severe neurological disorders, or any significant diseases affecting the gastrointestinal, cardiovascular, hepatic, renal, hematological, oncological, endocrine, respiratory, or immune systems, or other serious illnesses.
2. Diagnosis of claustrophobia.
3. History of drug abuse or alcohol dependence.
4. Pregnant or breastfeeding women.
5. Poor venous access that would preclude repeated venipuncture.
6. Use of experimental drugs or devices within one month prior to the study, where the safety or efficacy has not been established.
7. Any condition that the study investigators deem could pose potential harm or jeopardize participant safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety of Al18F-NOTA-Pentixafor | From radiotracer injection to 24 hours post-injection.
  Adverse effects were recorded according to CTCAE (version 5.0) after radiotracer injection and PET scan.
Diagnostic accuracy of Al18F-NOTA-Pentixafor PET/CT for PA | Through study completion, 1-1.5 years (from enrollment to to the final clinical or pathological diagnosis at 6-month follow-up after Al18F-NOTA-Pentixafor PET/CT )
  SUVmax and SUVmean of adrenal lesions, normal adrenal glands, and liver will be measured. The lesion-to-liver ratio (LLR) and lesion-to-normal adrenal ratio (LAR) will be calculated. Two nuclear medicine physicians will independently review the images, and a third physician will adjudicate in case of disagreement to reach a final diagnosis. Surgical pathology results or adrenal vein sampling (AVS) findings will serve as the reference standard to determine the sensitivity and specificity .
Surgical outcomes guided by Al18F-NOTA-Pentixafor PET/CT | Through study completion, 1-1.5 years (from enrollment to 6-month follow-up after surgery guided by Al18F-NOTA-Pentixafor PET/CT)
  Primary Aldosteronism Surgical Outcome (PASO) Criteria :
  1. Complete Clinical Success:Blood pressure is completely normalized without the need for antihypertensive medications.
  2. Partial Clinical Success:Blood pressure improves, requiring fewer antihypertensive medications or easier control.
  3. Absent Clinical Success:No significant improvement in blood pressure, and medication requirements remain unchanged.
  4. Complete Biochemical Success: Postoperative aldosterone-to-renin ratio normalizes, indicating full correction of aldosterone overproduction.
  5. Partial Biochemical Success: Aldosterone levels decrease but do not fully normalize.
  6. Absent Biochemical Success: No significant improvement in biochemical markers, suggesting persistent aldosterone overproduction.

SECONDARY OUTCOMES:
SUVmax of normal organs | From study completion to 6 months after completion.
  The biodistribution of Al18F-NOTA-Pentixafor will be assessed in the following organs: pituitary gland, parotid glands, thyroid glands, lungs, blood pool, liver, spleen, pancreas (including the head and uncinate process), gallbladder, stomach, small intestine, kidneys, and adrenal glands. The SUVmax values for these organs will be measured and documented.
Absorbed dose of target organs | From study completion to 6 months after completion.
  Absorbed dose of target organs were calculated using HERMES software.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China